CLINICAL TRIAL: NCT06404359
Title: Effects of a Strength Physical Exercise Program in Colorectal Cancer Patients Undergoing Chemotherapy Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juan Luis Sanchez Gonzalez (Other)
Responsible Party: Sponsor-Investigator, Juan Luis Sanchez Gonzalez, Principal Investigator. Dr. Juan Luis Sánchez González, University of Salamanca
Organization: University of Salamanca (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OncoExercise
Record Dates: First submitted 2024-04-30; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Oncology; Chemotherapy-induced Peripheral Neuropathy
Keywords: Exercise; Physiotherapy
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The investigators propose a 12-week intervention with therapeutic strength exercise in patients with colorectal cancer who are receiving chemotherapy treatment.
  Interventions: Other: Exercise
- Control group (Active Comparator): They will be provided with clear and concrete recommendations of activities for the user to perform the rest of the days of the week in order to increase their level of physical activity and increase weekly metabolic expenditure.
  Interventions: Other: Physical activity recommendations

INTERVENTIONS:
Other: Exercise — There will be 2 weekly sessions of 50 minutes, always guided by a physiotherapist, with the following distribution:
  1.- Warm-up: 15 minutes of global exercises of strength and resistance, focusing on the areas that are going to be worked as a priority in that session.
  Strength training: 6 to 8 strength exercises of large muscle groups. The approximate duration will be 25 minutes.
  3.- Cool down / cool down: Combination of breathing exercises and stretching, 10 minutes.
  Monitoring with activity bracelets.
  Arms: Exercise group
Other: Physical activity recommendations — They will be provided with a physical activity plan to be followed on a weekly basis.
  Arms: Control group

SUMMARY:
Chemotherapy is a crucial treatment in the fight against colon cancer, but unfortunately, its impact is not limited to cancer cells alone. Chemotherapy drugs, designed to attack fast-growing cells, also affect healthy tissues, leading to various side effects. One of the most common adverse effects is peripheral neuropathy, a condition that affects the peripheral nerves and can manifest as tingling sensations, numbness, pain or weakness in the extremities.

Chemotherapy-induced peripheral neuropathy can be especially challenging for colon cancer patients, as it further aggravates quality of life during an already difficult period. Nerves responsible for motor and sensory function are compromised, affecting the patient's ability to perform daily activities and weakening their physical endurance. This phenomenon adds to the emotional and physical burden of fighting cancer.

However, there are tools that can positively influence these adverse effects, such as physical exercise. Although it may seem contradictory, regular physical exercise has been shown to have beneficial effects on peripheral neuropathy. Physical exercise can improve blood circulation and promote regeneration of damaged peripheral nerves. In addition, exercise helps to alleviate the pain and discomfort associated with neuropathy, thereby strengthening patients' functional capacity.

It is essential to emphasize that any exercise plan must be tailored to the individual capabilities of each patient, and medical supervision is essential. Therefore, the combination of chemotherapy and carefully planned physical exercise offers a comprehensive strategy to address both the disease and its side effects, providing colon cancer patients with a better quality of life during their journey to recovery.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with colorectal cancer and who are receiving chemotherapy treatment.
* Sedentary people who have not performed physical activity in the last 8 weeks.
* Ability to understand the evaluation tests and the performance of the exercises.
* Presence of XXX symptoms (If we focus on neuropathy, it should be inclusion criteria).
* Voluntary participation in the study.

Exclusion Criteria:

- Present contraindication/s for physical exercise (musculoskeletal diseases, severe cardiovascular disease, bone metastases,...).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy-induced neuropathy | Baseline and immediately after the intervention
  The EORTC CIPN20 questionnaire will be used.This questionnaire contains 20 items on which patients rate their experience for each symptom during the previous week using scores from 1 (not at all) to 4 (very much). The sum score was obtained by adding the scores of items 1 to 19 resulting in a sum score range of 19 to 76, which was termed CIPN20 sum1-19. Item 20 rates male impotence

SECONDARY OUTCOMES:
Wellbeing | Baseline and immediately after the intervention
  It will be evaluated through the the EORTC QLG Core Questionnaire (EORTC QOL-30) quality of life questionnaire in its specific version for colorectal cancer EORT QLQ-CR30. Scores can range from 0 (worst quality of life) to 100 (best quality of life), with higher values indicating better quality of life in the areas evaluated.
Body Mass Index | Baseline and immediately after the intervention
  Obtained from the participant's weight and height.
Oxygen consumption | Before and after the intervention
  It will be evaluated through the 6-minute walk test.
Anxiety and depression | Baseline and immediately after the intervention
  They will be evaluated through the Hospital Anxiety and Depression Scale (HADS). Scores on the HADS can be interpreted as follows:
  Anxiety:
  0-7: Absence of clinically significant anxiety. 8-10: Possible presence of clinically significant anxiety. 11 or more: Clinically significant anxiety.
  Depression:
  0-7: Absence of clinically significant depression. 8-10: Possible presence of clinically significant depression. 11 or more: Clinically significant depression.
Fatigue | Baseline and immediately after the intervention
  The Functional Assessment of Cancer Therapy (FACT-F) Questionnaire will be used. FACT-F scores are calculated by summing the scores of the different domains, where higher scores indicate better quality of life. The total score may vary depending on the scale used in the specific questionnaire, but generally ranges from 0 to 176 points.
Sleep quality | Baseline and immediately after the intervention
  Will be evaluated through the Minimal Insomnia Symptom Scale (MISS). Each question is scored on a scale of 0 to 4, where 0 indicates that the symptom is not present and 4 indicates a very severe presence of the symptom. Therefore, the total score on the MISS can range from 0 to 12 points.
  Interpretations of the MISS scores may be as follows:
  0-3 points: Absence or minimal presence of insomnia symptoms. 4-6 points: Mild insomnia symptoms. 7-9 points: Moderate insomnia symptoms. 10-12 points: Severe insomnia symptoms.
Sex | Baseline
  It will be registered at the beginning of the study.
Heighth | Baseline
  It will be registered at the beginning of the study in centimeters.

IPD SHARING:
Plan to Share IPD: Undecided
Upon request by e-mail to the principal investigator